CLINICAL TRIAL: NCT00077116
Title: Idarubicin and Ara-C in Combination With Gemtuzumab-Ozogamicin (IAGO) for Young Untreated Patients, Without an HLA Identical Sibling, With High Risk MDS or AML Developing After a Preceding Period With MDS During 6 Months Duration: A Phase II Study
Brief Title: Idarubicin, Cytarabine, and Gemtuzumab Ozogamicin in Treating Patients With Previously Untreated High-Risk Myelodysplastic Syndrome or Acute Myeloid Leukemia Secondary to Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-06013; EORTC-06013
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: untreated adult acute myeloid leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Congenital Abnormalities | interventions — Busulfan; Cyclophosphamide; Cytarabine; Gemtuzumab; Idarubicin; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: cytarabine
Drug: gemtuzumab ozogamicin
Drug: idarubicin
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as gemtuzumab ozogamicin, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Giving monoclonal antibody therapy together with chemotherapy may kill more cancer cells. Giving healthy stem cells from a donor whose blood closely resembles the patient's blood will help the patient's bone marrow make new stem cells that become red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well giving idarubicin and cytarabine together with gemtuzumab ozogamicin works in treating patients with previously untreated high-risk myelodysplastic syndrome or acute myeloid leukemia secondary to myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of combining gemtuzumab ozogamicin with idarubicin and cytarabine with or without cyclophosphamide with total body irradiation vs busulfan followed by allogeneic stem cell transplantation in patients with previously untreated high-risk myelodysplastic syndromes (MDS) or acute myeloid leukemia secondary to MDS.
* Determine the toxicity profile of this regimen in these patients.
* Determine the antileukemic/anti-MDS activity of this regimen in these patients.

Secondary

* Determine the hepatotoxicity of this regimen, in terms of veno-occlusive disease, in these patients.
* Determine the severity of pancytopenia and duration of recovery in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 treatment groups.

* Group 1 (for patients with no HLA-matched sibling donor): Patients receive remission-induction chemotherapy comprising idarubicin IV over 5 minutes on days 1, 3, and 5; cytarabine IV continuously over 24 hours on days 1-10; and gemtuzumab ozogamicin IV over 2 hours on day 7. Treatment continues for a second course in the absence of unacceptable toxicity.
* Group 2 (for patients with an HLA-matched sibling donor): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive myeloablative consolidation chemotherapy comprising cyclophosphamide on days -6 and -5 and total body irradiation twice daily on days -4 to -2.
  * Arm II: Patients receive myeloablative consolidation chemotherapy comprising busulfan on days -8 to -5 and cyclophosphamide on days -4 and -3.

Patients in both arms may alternatively undergo T-cell depletion and/or a reduced-intensity conditioning regimen.

Approximately 4-8 weeks after completion of consolidation chemotherapy, all patients in group 2 undergo allogeneic bone marrow transplantation or allogeneic peripheral blood stem cell transplantation. Patients in group 2 then proceed to remission-induction chemotherapy as in group 1.

Patients achieving complete remission are recommended for consolidation therapy off study.

Patients are followed monthly for 6 months, every 2 months for 6 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study within 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * High-risk myelodysplastic syndromes (MDS), including any of the following:

    * Refractory anemia with excess blasts (RAEB) with > 10% blast cells in the bone marrow
    * RAEB in transformation
    * Other forms of MDS with multiple (3 or more) chromosomal abnormalities or chromosome 7 abnormalities AND/OR profound cytopenias, defined as neutrophil count < 500/mm^3 and/or platelet count < 20,000/mm^3
    * Chronic myelomonocytic leukemia with > 5% blast cells in the bone marrow
    * Chronic myelomonocytic leukemia with neutrophil count > 16,000/mm^3 OR monocyte count > 2,600/mm^3
  * Secondary acute myeloid leukemia supervening after overt MDS of more than 6 months in duration
* Patients with or without an HLA-identical sibling
* No active CNS leukemia

PATIENT CHARACTERISTICS:

Age

* 16 to 70

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No severe cardiovascular disease
* No arrhythmias requiring chronic treatment
* No congestive heart failure
* No symptomatic ischemic heart disease

Pulmonary

* No severe lung disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No HIV positivity
* No other concurrent malignant disease
* No active uncontrolled infection
* No history of alcohol abuse (i.e., averaged less than 5 alcoholic consumptions daily for the past year)
* No concurrent severe neurological or psychiatric disease
* No other psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 6 weeks since prior growth factors

Chemotherapy

* No prior intensive chemotherapy
* More than 6 weeks since prior low-dose chemotherapy or hydroxyurea

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 6 weeks since prior immunosuppressants
* No prior participation in this clinical study

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-11; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Rate of complete remission (CR) or complete remission with incomplete recovery of platelets (CRp) as measured by Cheson response criteria after the start of treatment
Severe toxicity after the start of treatment

SECONDARY OUTCOMES:
Disease-free survival from CR/CRp
Duration of overall survival
Severity of pancytopenia and duration of recovery in patients who reached CR/CRp after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Theo De Witte, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (9):
- Belgium (4):
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - H. Hartziekenhuis - Roeselaere., Roeselare
- Ruprecht - Karls - Universitaet Heidelberg, Heidelberg, Germany
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
- Universitaetsspital-Basel, Basel, Switzerland